CLINICAL TRIAL: NCT01410851
Title: The Acute Effects of Pulse Consumption on Glycaemic Responses and Measures of Satiety and Satiation
Brief Title: Pulses, Satiation, Food Intake and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: G. Harvey Anderson, Ph.D., Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PURENet:-Pulses and Satiation
Record Dates: First submitted 2011-07-27; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Pasta, tomato sauce & added chickpeas (Experimental): The pulse treatments and control (pasta with tomato sauce) were made the day before the session and the recipe was calculated to provide 1500 kcal at each session. All meals had the same energy density (~77kcal/100g). Calories derived from pulses were consistent among all pulse treatments (44%). The pulse treatments and control all contained macaroni pasta and homemade tomato sauce.
  Interventions: Other: dietary treatment
- Pasta, tomato sauce and added lentils (Experimental): The pulse treatments and control (pasta with tomato sauce) were made the day before the session and the recipe was calculated to provide 1500 kcal at each session. All meals had the same energy density (~77kcal/100g). Calories derived from pulses were consistent among all pulse treatments (44%). The pulse treatments and control all contained macaroni pasta and homemade tomato sauce.
  Interventions: Other: dietary treatment
- Pasta, tomato sauce and added navy beans (Experimental): The pulse treatments and control (pasta with tomato sauce) were made the day before the session and the recipe was calculated to provide 1500 kcal at each session. All meals had the same energy density (~77kcal/100g). Calories derived from pulses were consistent among all pulse treatments (44%). The pulse treatments and control all contained macaroni pasta and homemade tomato sauce.
  Interventions: Other: dietary treatment
- Pasta, tomato sauce with yellow peas (Experimental): The pulse treatments and control (pasta with tomato sauce) were made the day before the session and the recipe was calculated to provide 1500 kcal at each session. All meals had the same energy density (~77kcal/100g). Calories derived from pulses were consistent among all pulse treatments (44%). The pulse treatments and control all contained macaroni pasta and homemade tomato sauce.
  Interventions: Other: dietary treatment
- Pasta and tomato sauce (Experimental): The pulse treatments and control (pasta with tomato sauce) were made the day before the session and the recipe was calculated to provide 1500 kcal at each session. All meals had the same energy density (~77kcal/100g). Calories derived from pulses were consistent among all pulse treatments (44%). The pulse treatments and control all contained macaroni pasta and homemade tomato sauce.
  Interventions: Other: dietary treatment

INTERVENTIONS:
Other: dietary treatment — A within-subject, balanced repeated-measures design was followed where subjects received 4 treatments or control over 5 weeks approximately 1 week apart. The pulse treatments contained: (1) chickpeas (Primo, Toronto, ON), (2) lentils (Primo, Toronto, ON), (3) navy beans (Ferma, Toronto, ON) or (4) yellow peas (Nupak, Toronto, ON).

SUMMARY:
Pulses have the potential to be positioned as a food for body weight and metabolic control based on their composition, effects on rate of digestion and absorption of fat and carbohydrates, and effects on satiety. However, the role of individual pulses incorporated into a mixed meal on regulation of food intake, satiety and glycaemic control remains unclear. Therefore, the objective of our study was to determine the effects of ad libitum consumption of pulse meals (treatments) on food intake at an ad libitum pulse meal, food intake at an ad libitum pizza meal at four hours, subjective appetite and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young males with BMI of 20-24.9 kg/m2

Exclusion Criteria:

* Females
* Smokers
* Breakfast skippers
* Individuals with diabetes or other metabolic diseases
* Those scoring ≥ 11 on an Eating Habit Questionnaire

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Short-term energy intake | over 280 min
  Energy intake was measured at the treatment meal (0-20 min) and at a pizza meal (second meal) provided four hours later (260-280 min).

SECONDARY OUTCOMES:
Blood glucose and satiety | 20, 40, 60, 110, 140, 200, 260, 280, 300, 320 and 340 min
  Following treatment meal consumption, blood glucose and appetite were measured at 20, 40, 60, 110, 140, 200 and 260 min and are reported as pre-second meal values. Following the pizza meal, blood glucose and appetite were measured at 280, 300, 320 and 340 min and are reported as post-second meal values.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada